CLINICAL TRIAL: NCT00172237
Title: Proprioception and Eye-head Coordination for the Cervical Spine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Shwu-Fen Wang/Professor, Department and Graduate School of Physical Therapy, National Taiwan University
Other Study IDs: 5460
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2010-01

CONDITIONS: Spinal Diseases
Keywords: eye-head coordination; proprioception; cervical spine with degenerative disease; degenerated cervical spine
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Specific aims of this project were as follows:

1. To investigate the eye-head coordination of patients with cervical spine degeneration.
2. To investigate the relationship of these impairment measurements (range of motion, muscle power, proprioception, sensory threshold, eye-head coordination) and functional outcome (neck disability index, quality of life evaluation).
3. To develop a computer assistant device and software for the proprioceptive training and eye-head coordination.
4. To provide a treatment and prevention program emphasized on proprioception treatment and coordination for employee with neck-shoulder complaints.

ELIGIBILITY:
Inclusion Criteria:

* Group one: participants without degenerated disease in cervical spine
* Group two: participants with degenerated disease in cervical spine

Exclusion Criteria:

* Grade III, IV degenerated cervical spine

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 45-64 year-old healthy adults and adults with neck pain
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-12; Study Completion 2010-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shwu-Fen Wang, Ph.D, Study Chair — School and Graduate Institute of Physical Therapy, National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy, Taipei, Taiwan